CLINICAL TRIAL: NCT04162886
Title: Effects of Thrower's Ten Exercises on Upper Extremity Strength, Power and Balance
Brief Title: Effects of Exercises on Physical Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Özge Gökalp, Principal Investigator, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017/45-03
Record Dates: First submitted 2019-11-12; First posted 2019-11-14 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Physical Performance
Keywords: Exercise; power; muscle strength; balance
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Thrower's ten exercises will given for 8 weeks, 3 days in a week.
  Interventions: Other: Exercise
- Control Group (No Intervention): Nothing given to the control group, will be told to continue their normal life for 8 weeks.

INTERVENTIONS:
Other: Exercise — Thrower's ten exercises will given for 8 weeks, 3 days in a week.
  Arms: Exercise Group

SUMMARY:
Aim: The aim of the study was to investigate the effects of thrower's ten exercises on the upper extremity performance in healthy sedentary individuals.

Method: 36 healthy sedentary men and women aged 18-35 years will be included in the study. Subjects will be divided into two groups: exercise and control. The exercise group will be given Thrower's Ten training sessions 3 times a week over an 8-week period. Before and after the study, the subjects were tested for dynamic balance on the upper extremity with the Upper Limp Y balance test and for explosive power with the medicine ball throw test. Moreover, the strength of the shoulder rotator muscles was measured with an isokinetic dynamometer at a speed of 60º/sec.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women and men aged 18-35 years

Exclusion Criteria:

* Individuals with any neurological, orthopedic, cardiovascular, psychological problems,
* individuals who have a musculoskeletal injury in the last 1 year,
* individuals who doing regular physical activity/sport in the last 6 months

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-29 (Actual)

PRIMARY OUTCOMES:
Change in the level of upper extremity strength assessed by an isokinetic dynamometer (Cybex Norm). | At the beginning and at the end of 8 weeks.
  During all tests, participants will be encouraged verbally and visually. The forces of the upper extremity will be measured with an isokinetic dynamometer and an angular velocity of 5 repetitions at 60 ° / sec. Before the actual exam, subjects will allowed to make 3 trials. The test results will be recorded for the dominant side.

SECONDARY OUTCOMES:
Change in the level of upper extremity explosive strength assessed by a seated medicine ball throw (SMBT) test. | At the beginning and at the end of 8 weeks.
  A line will be drawn on a flat surface before testing. In the beginning, the subject will sits on this line with the head, back, and butt leaning against the wall and legs extending straight following the line. Hands were placed on the two sides of the wall without fingers touching. Upon the start command, the subject will lifted the ball to the chest and threw forwards as in a basketball shot. A 2 kg medicine ball will used in the test.

OTHER OUTCOMES:
Change in the level of upper extremity balance assessed using Upper Quarter Y Balance Test (UQYBT) | At the beginning and at the end of 8 weeks.
  Participants will put the dominant or non-dominant hand to be tested on the starting line and extended the arm in medial, inferior lateral, and superior lateral directions and the length will measured in all 3 directions in cm.

CONTACTS AND LOCATIONS:
Overall Officials: Berkiye Kırmızıgil, Asst. Prof, Study Chair — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gokalp O, Kirmizigil B. Effects of Thrower's Ten exercises on upper extremity performance: A randomized controlled study. Medicine (Baltimore). 2020 Oct 16;99(42):e22837. doi: 10.1097/MD.0000000000022837. PMID 33080765